CLINICAL TRIAL: NCT01964989
Title: A Phase III, Stratified, Randomized, Observer Blind, Controlled, Multicenter Clinical Study to Evaluate the Safety, Immunogenicity and Efficacy of an Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine Compared to Non-Adjuvanted Comparator Influenza Vaccine in Children ≥6 to < 72 Months of Age.
Brief Title: Clinical Study to Evaluate the Safety, Immunogenicity and Efficacy of Investigational Flu Vaccine Compared to Approved Flu Vaccine in Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V118_05; 2012-000218-12 (EudraCT Number)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Influenza Virus
Keywords: Influenza; children
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aQIV (Experimental): flu vaccine
  Interventions: Biological: Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV)
- non-adjuvanted comparator (Active Comparator): flu vaccine
  Interventions: Biological: Non-adjuvanted Trivalent Influenza Vaccine (TIV) / Quadrivalent Influenza Vaccine (QIV)

INTERVENTIONS:
Biological: Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine (aQIV) — 1 or 2 doses (naïve / non-naive subjects) 0.25 ml: ≥6 months to <36 months, 0.5 ml: ≥36 months to <72 months
  Arms: aQIV
Biological: Non-adjuvanted Trivalent Influenza Vaccine (TIV) / Quadrivalent Influenza Vaccine (QIV) — 1 or 2 doses (naïve / non-naive subjects) 0.25 ml: ≥6 months to <36 months, 0.5 ml: ≥36 months to <72 months
  Arms: non-adjuvanted comparator

SUMMARY:
Safety, Immunogenicity and Efficacy of an Adjuvanted Quadrivalent Subunit Influenza Virus Vaccine Compared to Non-Adjuvanted Comparator Influenza Vaccine in Children ≥6 to <72 Months of Age. The study was conducted during the 2013/2014 and 2014/2015 northern hemisphere influenza season.

ELIGIBILITY:
Inclusion Criteria:

* Children, males and females, healthy or at high risk of complications from influenza, between ≥6 months to <72 months of age
* Documented consent provided by the subject's parent(s)/legal guardian(s)
* Subjects and/or subject's parent(s)/legal guardian(s) able to comply with all study procedures.

Exclusion Criteria:

* Children with history of allergy to vaccine components.
* Additional eligibility criteria may be discussed by contacting the site

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10644 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Seqirus
Locations (167):
- United States (91):
  - 222, Novartis Investigational Site, Chandler, Arizona
  - 267, Novartis Investigational Site, Harrisburg, Arkansas
  - 259, Novartis Investigational Site, Anaheim, California
  - 280, Novartis Investigational Site, Anaheim, California
  - 213, Novartis Investigational Site, Baldwin Park, California
  - 407, Novartis Investigational Site, Downey, California
  - 238, Novartis Investigational Site, La Puente, California
  - 411, Novartis Investigational Site, Ontario, California
  - 202, Novartis Investigational Site, Paramount, California
  - 250, Novartis Investigational Site, San Diego, California
  - 293, Novartis Investigational Site, San Francisco, California
  - 243, Novartis Investigational Site, Colorado Springs, Colorado
  - 249, Novartis Investigational Site, Denver, Colorado
  - 229, Novartis Investigational Site, Boca Raton, Florida
  - 416, Novartis Investigational Site, Hialeah, Florida
  - 287, Novartis Investigational Site, Hialeah, Florida
  - 412, Novartis Investigational Site, Homestead, Florida
  - 224, Novartis Investigational Site, Melbourne, Florida
  - 417, Novartis Investigational Site, Miami, Florida
  - 404, Novartis Investigational Site, Miami, Florida
  - 285, Novartis Investigational Site, Miami, Florida
  - 277,Novartis Investigational Site, Miami, Florida
  - 234, Novartis Investigational Site, Opa-locka, Florida
  - 297, Novartis Investigational Site, Orlando, Florida
  - 297, Novartis Investigational vaccine, Orlando, Florida
  - 410, Novartis Investigational Site, Sarasota, Florida
  - 401, Novartis iNvestiagtional Site, Atlanta, Georgia
  - 299, Novartis Investigational Site, DeKalb, Illinois
  - 268, Novartis Investigational Site, Peoria, Illinois
  - 209, Novartis Investigational Site, Augusta, Kansas
  - 210, Novartis Investigational Site, Newton, Kansas
  - 274 Novartis Investigational Site, Park City, Kansas
  - 211, Novartis Investigational Site, Wichita, Kansas
  - 269, Novartis Investigational Site, Bardstown, Kentucky
  - 226, Novartis Investigational Site, Louisville, Kentucky
  - 248, Novartis Investigational Site, Louisville, Kentucky
  - 207, Novartis Investigational Site, Louisville, Kentucky
  - 290, Novartis Investigational Site, Louisville, Kentucky
  - 265, Novartis Investigational Site, Haughton, Louisiana
  - 408, Novartis Investigational Site, Mangham, Louisiana
  - 225, Novartis Investigational Site, Metairie, Louisiana
  - 233, Novartis Investigational Site, Metairie, Louisiana
  - 418, Novartis Investigational SIte, Monroe, Louisiana
  - 262, Novartis Investigational site, Annapolis, Maryland
  - 263, Novartis Investigational Site, Frederick, Maryland
  - 405, Novartis Investigational Site, Silver Spring, Maryland
  - 278, Novartis Investigational Site, Saint Paul, Minnesota
  - 221, Novartis Investigational Site, Bellevue, Nebraska
  - 219, Novartis Investigational Site, Fremont, Nebraska
  - 402, Novartis Investigational Site, Omaha, Nebraska
  - 288, Novartis Investigational Site, Omaha, Nebraska
  - 228, Novartis Investigational Site, Omaha, Nebraska
  - 244, Novartis Investigational Site, Henderson, Nevada
  - 286, Novartis Investigational site, Las Vegas, Nevada
  - 255, Novartis Investigational Site, Binghamton, New York
  - 414, Novartis Investigational Site, Brooklyn, New York
  - 264, Novartis Investigational Site, Syracuse, New York
  - 409, Novartis Investigational Site, Boone, North Carolina
  - 266, Novartis Investigational Site, Cary, North Carolina
  - 403, Novartis Investigational Site, Clyde, North Carolina
  - 240, Novartis Investigational Site, Akron, Ohio
  - 254, Novartis Investigational Site, Cleveland, Ohio
  - 245, Novartis Investigational Site, Dayton, Ohio
  - 281, Novartis Investigational Site, Dayton, Ohio
  - 281, Novartis Investigational vaccines, Dayton, Ohio
  - 256, Novartis Investigational Site, Tulsa, Oklahoma
  - 292, Novartis Investigational Site, Erie, Pennsylvania
  - 270, Novartis Investigational Site, Scottdale, Pennsylvania
  - 220, Novartis Investigational Site, Anderson, South Carolina
  - 406, novartis Investigational Site, Barnwell, South Carolina
  - 272, Novartis Investigational Site, Charleston, South Carolina
  - 232, Novartis Investigational Site, Moncks Corner, South Carolina
  - 291, Novartis Investigational vaccine, Spartanburg, South Carolina
  - 283, Novartis Investigational Site, Nashville, Tennessee
  - 208, Novartis Investigational Site, Austin, Texas
  - 247, Novartis Investigational Site, Fort Worth, Texas
  - 217, Novartis Investigational Site, Fort Worth, Texas
  - 214, Novartis Investigational Site, San Angelo, Texas
  - 400, Novartis investigational Site, San Antonio, Texas
  - 260, Novartis Investigational Site, Tomball, Texas
  - 295, Novartis Investigational Site, Layton, Utah
  - 236, Novartis Investigational Site, Salt Lake City, Utah
  - 212, Novartis Investigational Site, Salt Lake City, Utah
  - 246, Novartis Investigational Site, Salt Lake City, Utah
  - 279, Novartis Investigational Site, Spanish Fork, Utah
  - 282, Novartis Investigational Site, Syracuse, Utah
  - 294, Novartis Investigational Site, West Haven, Utah
  - 201, Novartis Investigational Site, West Jordan, Utah
  - 271, Novartis Investigational Site, West Jordan, Utah
  - 251, Novartis Investigational Site, Burke, Virginia
  - 296, Novartis Investigational Site, Vienna, Virginia
- Canada (5):
  - 184, Novartis Investigational Site, Greater Sudbury, Ontario
  - 180, Novartis Investigational Site, Newmarket, Ontario
  - 182,Novartis Investigational Site, Toronto, Ontario
  - 183, Novartis Investigational Site, Québec
  - 186, Novartis Investigational Site, Québec
- Finland (11):
  - 001, Novartis Investigational Site, Espoo
  - 003, Novartis Investigational Site, Helsinki
  - 002, Novartis Investigational Site, Helsinki
  - 004, Novartis Investigational Site, Jarvenpaa
  - 005, Novartis Investigational Site, Kokkola
  - 006, Novartis Investigational Site, Oulu
  - 007, Novartis Investigational Site, Pori
  - 008, Novartis Investigational Site, Seinäjoki
  - 009, Novartis Investigational Site, Tampere
  - 010, Novartis Investigational Site, Turku
  - 011, Novartis Investigational Site, Vantaa
- Italy (9):
  - 030, Novartis Investigational Site, Florence
  - 023, Novartis Investigational Site, Genova
  - 020, Novartis Investigational Site, Milan
  - 026, Novartis Investigational Site, Milan
  - 025, Novartis Investigational Site, Napoli
  - 021, Novartis Investigational Site, Novara
  - 022, Novartis Investigational Site, Padua
  - 024, Novartis Investigational Site, Pisa
  - 028, Novartis Investigational Site, Sassari
- Mexico (6):
  - 173, Novartis Investigational Site, Morelia, Michoacán
  - 176, Novartis Investigational Site, Durango
  - 170, Novartis Investigational Site, México
  - 177, Novartis Investigational Site, México
  - 178, Novartis Investigational Site, México
  - 175, Novartis Investigational Site, México
- Philippines (7):
  - 300, Novartis Investigational Site, Dasmariñas, Cavite
  - 306, Novartis Investigational Site, Alabang, Muntilupa
  - 303, Novartis Investigational Site, City of Muntinlupa
  - 304, Novartis Investigational Site, City of Muntinlupa
  - 305, Novartis Investigational Site, City of Muntinlupa
  - 302, Novartis Investigational Site, Manila
  - 301, Novartis Investigational Site, Manila
- Poland (13):
  - 040, Novartis Investigational Site, Dębica
  - 042, Novartis Investigational Site, Katowice
  - 048, Novartis Investigational Site, Lodz
  - 049, Novartis Investigational Site, Lubartów
  - 051, Novartis Investigational Site, Oborniki Śląskie
  - 046, Novartis Investigational Site, Osielsko
  - 043, Novartis Investigational Site, Siemianowice Śląskie
  - 047, Novartis Investigational Site, Tarnów
  - 041, Novartis Investigational Site, Warsaw
  - 050, Novartis Investigational Site, Warsaw
  - 045, Novartis Investigational Site, Wola
  - 044, Novartis Investigational Site, Wroclaw
  - 052, Novartis Investigational Site, Łęczna
- Puerto Rico (3):
  - 257, Novartis Investigational Site, Ponce
  - 415, Novartis Investigational vaccine, San Juan
  - 415, Novartis Investigational Site, San Juan
- Spain (7):
  - 80, Novartis Investigational Site, Sabadell, Barcelona
  - 075, Novartis Investigational Site, Santiago de Compostela, Galicia
  - 074, Novartis Investigational Site, Granada
  - 076, Novartis Investigational Site, Madrid
  - 077, Novartis Investigational Site, Madrid
  - 79, Novartis Investigational Site, Málaga
  - 078, Novartis Investigational Site, Valencia
- Taiwan (7):
  - 343, Novartis Investigational Site, Banqiao District, New Taipei City
  - 346, Novartis Investigational Site, Datong, Taipei City
  - 344, Novartis Investigational Site, Taichung
  - 345, Novartis Investigational Site, Taichung
  - 340, Novartis Investigational Site, Taipei
  - 341, Novartis Investigational Site, Taipei
  - 342, Novartis Investigational Site, Taoyuan District
- Thailand (8):
  - 321, Novartis Investigational Site, Bangkoknoi, Bangkok
  - 322, Novartis Investigational Site, Bangkoknoi, Bangkok
  - 323, Novartis Investigational Site, Pathum Wan, Bangkok
  - 327, Novartis Investigational Site, Ratchathewi, Bangkok
  - 325, Novartis Investigational Site, Pathum Thani, Changwat Pathum Thani
  - 326, Novartis Investigational Site, Hat Yai, Songkhia
  - 320, Novartis Investigational Site, Bangkok
  - 324, Novartis Investigational Site, Bangkok

REFERENCES:
- [Derived] Esposito S, Fling J, Chokephaibulkit K, de Bruijn M, Oberye J, Zhang B, Vossen J, Heijnen E, Smolenov I. Immunogenicity and Safety of an MF59-adjuvanted Quadrivalent Seasonal Influenza Vaccine in Young Children at High Risk of Influenza-associated Complications: A Phase III, Randomized, Observer-blind, Multicenter Clinical Trial. Pediatr Infect Dis J. 2020 Aug;39(8):e185-e191. doi: 10.1097/INF.0000000000002727. PMID 32404782
- [Derived] Vesikari T, Kirstein J, Devota Go G, Leav B, Ruzycky ME, Isakov L, de Bruijn M, Oberye J, Heijnen E. Efficacy, immunogenicity, and safety evaluation of an MF59-adjuvanted quadrivalent influenza virus vaccine compared with non-adjuvanted influenza vaccine in children: a multicentre, randomised controlled, observer-blinded, phase 3 trial. Lancet Respir Med. 2018 May;6(5):345-356. doi: 10.1016/S2213-2600(18)30108-5. Epub 2018 Apr 6. PMID 29631857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 146 sites in 9 countries.
Pre-assignment Details: All enrolled subjects were included in the trial. Non-naive participants received 1 dose of vaccine on Day 1 only. Naive participants received 2 doses of vaccine, the first dose on Day 1 and the second dose on Day 29.
Groups:
- aQIV (≥6 to <72 Months): Subjects ≥6 to <72 months of age who received aQIV
- TIV/QIV (≥6 to <72 Months): Subjects ≥6 to <72 months of age who received TIV/QIV
Period: Overall Study
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Started | 5352 | 5292
Completed | 4568 | 4545
Not Completed | 784 | 747
Not completed — Protocol Violation | 3 | 4
Not completed — Administrative Reason | 103 | 95
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 3
Not completed — Withdrawal by Subject | 156 | 160
Not completed — Lost to Follow-up | 254 | 232
Not completed — Other | 267 | 252

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months) | Total
Number analyzed (Participants) | 5352 | 5292 | 10644
Age, Continuous [Mean (Standard Deviation); unit: months] | 38.4 (18.43) | 38 (18.40) | 38.2 (18.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2643 | 2590 | 5233
  Male | 2709 | 2702 | 5411
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 664 | 632 | 1296
  Not Hispanic or Latino | 4678 | 4647 | 9325
  Unknown or Not Reported | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 11 | 21
  Asian | 2348 | 2361 | 4709
  Native Hawaiian or Other Pacific Islander | 14 | 16 | 30
  Black or African American | 711 | 692 | 1403
  White | 2153 | 2091 | 4244
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 116 | 121 | 237
Naivety Status [Count of Participants; unit: Participants]
  Vaccine Naive | 3611 | 3597 | 7208
  Vaccine Non-Naive | 1741 | 1695 | 3436

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint: First-Occurrence Reverse Transcription-Polymerase Chain Reaction (RT-PCR) Confirmed Influenza A and/or B of Any Influenza Strain in Subjects ≥6 to <72 Months of Age
Description: Relative efficacy of aQIV compared to non-adjuvanted comparator (TIV/QIV) was determined by the number of subjects ≥6 to <72 months of age with RT-PCR confirmed occurrence of influenza A and/or B of any influenza strain that occurred at ≥21 days and ≤180 days after the last vaccination or until the end of the influenza season, whichever was longer. Efficacy was determined on influenza cases caused by any of the influenza strains related to the two A subtypes and the B lineage(s) common to aQIV and TIV (i.e. A/H1N1, A/H3N2 and B/Yamagata during first influenza season), and common to aQIV and QIV (i.e. A/H1N1, A/H3N2 and both B lineages during second season and through the end of the trial).
Time Frame: ≥21 days and ≤180 days after the last vaccination or until the end of the influenza season (Northern Hemisphere: end of June; Southern Hemisphere: end of December; Philippines/Thailand: end of October), whichever was longer
Population: The Full Analysis Set for Efficacy consisting of all enrolled subjects who actually received a study vaccination and were evaluated for efficacy at least 21 days after the last vaccination was used for analysis.
Measure: Number; unit: Number of cases
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 5278 | 5193
Number of cases
  Any strain | 256 | 252
  A/H1N1 | 7 | 17
  A/H3N2 | 200 | 196
  B/Yamagata | 36 | 36
  B/Victoria | 14 | 9
Statistical Analysis 1: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Test type: Superiority — Relative vaccine efficacy (rVE; ≥6 to <72 months) rVE = (1-HR) is the relative vaccine efficacy of aQIV and HR is defined as hazard ratio between aQIV and non adjuvanted comparator; Cox Proportional Hazard = -0.67, 95% CI 2-sided [-19.81 to 15.41]

2. Secondary Outcome: Efficacy Endpoint: First-Occurrence RT-PCR Confirmed Influenza A and/or B of Any Influenza Strain in Subjects ≥6 to <24 Months, ≥6 to <36 Months and ≥36 to <72 Months of Age.
Description: Relative efficacy of aQIV compared to non-adjuvanted comparator (TIV/QIV) was determined by the number of subjects with RT-PCR confirmed occurrence of influenza A and/or B of any influenza strain that occurred at ≥21 days and ≤180 days after the last vaccination or until the end of the influenza season, whichever was longer. Efficacy was determined on influenza cases caused by any of the influenza strains related to the two A subtypes and the B lineage(s) common to aQIV and TIV (i.e. A/H1N1, A/H3N2 and B/Yamagata during first influenza season), and common to aQIV and QIV (i.e. A/H1N1, A/H3N2 and both B lineages during second season and through the end of the trial).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Number of cases
Groups:
- aQIV (≥6 to <24 Months): Subjects ≥6 to <24 months of age who received aQIV
- TIV/QIV (≥6 to <24 Months): Subjects ≥6 to <24 months of age who received TIV/QIV
- aQIV (≥6 to <36 Months): Subjects ≥6 to <36 months of age who received aQIV
- TIV/QIV (≥6 to <36 Months): Subjects ≥6 to <36 months of age who received TIV/QIV
- aQIV (≥36 to <72 Months): Subjects ≥36 to <72 months of age who received aQIV
- TIV/QIV (≥36 to <72 Months): Subjects ≥36 to <72 months of age who received TIV/QIV
Arm/Group | aQIV (≥6 to <24 Months) | TIV/QIV (≥6 to <24 Months) | aQIV (≥6 to <36 Months) | TIV/QIV (≥6 to <36 Months) | aQIV (≥36 to <72 Months) | TIV/QIV (≥36 to <72 Months)
Number analyzed (Participants) | 1299 | 1339 | 2484 | 2471 | 2794 | 2722
Number of cases
  Any Strain | 55 | 79 | 115 | 119 | 141 | 133
  A/H1N1 | 2 | 5 | 5 | 8 | 2 | 9
  A/H3N2 | 44 | 66 | 92 | 99 | 108 | 97
  B/Yamagata | 5 | 9 | 13 | 12 | 23 | 24
  B/Victoria | 4 | 0 | 5 | 1 | 9 | 8

3. Secondary Outcome: Efficacy Endpoint: First-Occurrence Culture Confirmed Influenza A and/or B of Any Influenza Strain in Subjects ≥6 to <72 Months, ≥6 to <24 Months, ≥6 to <36 Months and ≥36 to <72 Months of Age
Description: Relative efficacy of aQIV compared to non-adjuvanted comparator (TIV/QIV) was determined by the number of subjects with culture confirmed occurrence of influenza A and/or B of any influenza strain that occurred at ≥21 days and ≤180 days after the last vaccination or until the end of the influenza season, whichever was longer. Efficacy was determined on influenza cases caused by any of the influenza strains related to the two A subtypes and the B lineage(s) common to aQIV and TIV (i.e. A/H1N1, A/H3N2 and B/Yamagata during first influenza season), and common to aQIV and QIV (i.e. A/H1N1, A/H3N2 and both B lineages during second season and through the end of the trial).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months) | aQIV (≥6 to <24 Months) | TIV/QIV (≥6 to <24 Months) | aQIV (≥6 to <36 Months) | TIV/QIV (≥6 to <36 Months) | aQIV (≥36 to <72 Months) | TIV/QIV (≥36 to <72 Months)
Number analyzed (Participants) | 5278 | 5193 | 1299 | 1339 | 2484 | 2471 | 2794 | 2722
Number of cases
  Any strain | 140 | 146 | 31 | 48 | 64 | 68 | 76 | 78
  Matched strain | 74 | 80 | 19 | 32 | 35 | 42 | 39 | 38
  Unmatched strain | 65 | 62 | 12 | 14 | 29 | 23 | 36 | 39

4. Secondary Outcome: Efficacy Endpoint: First-occurrence RT-PCR and Culture Confirmed Influenza A and/or B of Any Influenza Strain in Subjects at High Risk of Influenza Complications
Description: Relative efficacy of aQIV compared to non-adjuvanted comparator (TIV/QIV) was determined by the number of subjects ≥6 to <72 months of age with RT-PCR confirmed and culture confirmed occurrence of influenza A and/or B of any influenza strain that occurred at ≥21 days and ≤180 days after the last vaccination or until the end of the influenza season, whichever was longer, in healthy subjects and subjects at risk of influenza related complications. Efficacy was determined on influenza cases caused by any of the influenza strains related to the two A subtypes and the B lineage(s) common to aQIV and TIV (i.e. A/H1N1, A/H3N2 and B/Yamagata during first influenza season), and common to aQIV and QIV (i.e. A/H1N1, A/H3N2 and both B lineages during second season and through the end of the trial).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Number of cases
Groups:
- aQIV (≥6 to <72 Months): Subjects ≥6 to <72 months of age who received aQIV: Healthy and at-risk
- TIV/QIV (≥6 to <72 Months): Subjects ≥6 to <72 months of age who received TIV/QIV: Healthy and at-risk
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 5278 | 5193
Number of cases
  Healthy RT-PCR: number analyzed (Participants) | 4819 | 4756
  Healthy RT-PCR | 244 | 233
  High Risk RT-PCR: number analyzed (Participants) | 459 | 437
  High Risk RT-PCR | 12 | 19
  Healthy Culture-confirmed: number analyzed (Participants) | 4819 | 4756
  Healthy Culture-confirmed | 130 | 136
  High Risk Culture-confirmed: number analyzed (Participants) | 459 | 437
  High Risk Culture-confirmed | 10 | 10

5. Secondary Outcome: Efficacy Endpoint: First-occurrence RT-PCR and Culture Confirmed Influenza A and/or B of Any Influenza Strain in Naive and Non-naive Subjects Separately
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Number of cases
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 5278 | 5193
Number of cases
  Vaccine Naive RT-PCR: number analyzed (Participants) | 3553 | 3525
  Vaccine Naive RT-PCR | 160 | 170
  Vaccine Non-naive RT-PCR: number analyzed (Participants) | 1725 | 1668
  Vaccine Non-naive RT-PCR | 96 | 82
  Vaccine Naive Culture-confirmed: number analyzed (Participants) | 3553 | 3525
  Vaccine Naive Culture-confirmed | 80 | 101
  Vaccine Non-naive Culture-confirmed: number analyzed (Participants) | 1725 | 1668
  Vaccine Non-naive Culture-confirmed | 60 | 45

6. Secondary Outcome: Efficacy Endpoint: First-occurrence RT-PCR-confirmed Influenza A and/or B of Any Influenza Strain in Subjects ≥6 to <72 Months of Age at ≥7 Days and at ≥14 Days After First Vaccination up to the Day of Second Vaccination in Vaccine naïve Subjects Only
Description: Relative efficacy of aQIV compared to non-adjuvanted comparator (TIV/QIV) was based on the number of vaccine naive subjects ≥6 to <72 months of age with RT-PCR confirmed occurrence of influenza A and/or B of any influenza strain that occurred at ≥7 days and ≥14 days after the first vaccination up to the day of the second vaccination. TIV was used as the comparator in Season 1; and QIV was used as the comparator in Season 2. Efficacy was determined on influenza cases caused by any of the influenza strains related to the two A subtypes and the B lineage(s) common to aQIV and TIV (i.e. A/H1N1, A/H3N2 and B/Yamagata during first influenza season), and common to aQIV and QIV (i.e. A/H1N1, A/H3N2 and both B lineages during second season and through the end of the trial).
Time Frame: ≥7 days and at ≥14 days after first vaccination up to day of second vaccination
Population: Full Analysis Set Early Efficacy: All subjects in the Enrolled Set who actually received a study vaccination and were evaluated for efficacy at least 7 days after the last vaccination.
Measure: Number; unit: Number of cases
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 3559 | 3535
Number of cases
  ≥7 days after first and up to second vaccination | 16 | 35
  ≥14 days after first and up to second vaccination | 8 | 27

7. Secondary Outcome: Efficacy Endpoint: First-occurrence RT-PCR-confirmed Influenza A and/or B of Any Influenza Strain in Subjects ≥6 to <72 Months of Age Occurring at ≥7 Days and ≤21 Days After Last Vaccination, in All Subjects.
Description: Relative efficacy of aQIV compared to non-adjuvanted comparator (TIV/QIV) was based on the number of vaccine naïve subjects ≥6 to <72 months of age with RT-PCR confirmed occurrence of influenza A and/or B of any influenza strain that occurred at ≥7 days and ≤21 after the last vaccination. TIV was used as the comparator in Season 1; and QIV was used as the comparator in Season 2. Efficacy was determined on influenza cases caused by any of the influenza strains related to the two A subtypes and the B lineage(s) common to aQIV and TIV (i.e. A/H1N1, A/H3N2 and B/Yamagata during first influenza season), and common to aQIV and QIV (i.e. A/H1N1, A/H3N2 and both B lineages during second season and through the end of the trial).
Time Frame: ≥7 days and ≤21 days after the last vaccination
Population: as for outcome 6
Measure: Number; unit: Number of cases
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 5286 | 5208
Number of cases | 4 | 15

8. Secondary Outcome: Immunogenicity Endpoint: Hemagglutination Inhibition (HI) Antibody Responses to aQIV vs TIV/QIV Against Each of the Vaccine Strains in Terms of Geometric Mean Titers (GMTs) and GMT Ratios in Subjects ≥6 to <72 Months of Age
Description: Pooled GMT values across both naïve and non-naïve subjects are provided for the Day 22/50 (ie, 21 days after last vaccination) and Day 181/209 (ie, 180 days after last vaccination) assessments; Nonadjuvanted TIV administered in Season 1 and nonadjuvanted QIV administered in Season 2; Homologous strains: A/H1N1=A/California/7/2009 pdm09-like virus, A/H3N2=A/Texas/50/2012, B/ Yamagata=B/Massachusetts/2/2012 and B/Victoria=B/Brisbane/60/2008; For B/Victoria results from Season 2 only are presented for both vaccine groups and used in the vaccine comparison analysis.
Time Frame: Baseline (Day 1), Day 29, Day 50 and Day 209 for vaccine naïve subjects; Baseline (Day 1), Day 22 and Day 181 for vaccine non-naïve subjects
Population: The Full Analysis Set for Immunogenicity consisting of all enrolled/randomized subjects who received a study vaccination AND provided evaluable serum samples (immunogenicity) for both before (baseline) and after vaccination was used for analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 1481 | 1405
titer
  A/H1N1, Day 1 | 40.08 [32.3 to 49.7] | 39.49 [31.8 to 49.1]
  A/H1N1, D22/50 | 996.40 [888.4 to 1117.6] | 522.50 [465.3 to 586.7]
  A/H1N1, D181/209 | 351.59 [311.2 to 397.2] | 189.43 [167.4 to 214.3]
  A/H3N2, Day 1 | 72.96 [58.1 to 91.6] | 70.38 [55.9 to 88.5]
  A/H3N2, D22/50 | 1153.4 [1035.4 to 1284.9] | 674.01 [604.4 to 751.6]
  A/H3N2, D181/209 | 458.07 [403.0 to 520.6] | 290.88 [255.5 to 331.1]
  B/Yamagata, Day 1 | 10.17 [9.0 to 11.5] | 10.12 [9.0 to 11.4]
  B/Yamagata, Day 22/50 | 198.89 [173.1 to 228.5] | 90.68 [78.8 to 104.3]
  B/Yamagata, Day 181/209 | 48.65 [42.9 to 55.2] | 26.22 [23.1 to 29.8]
  B/Victoria, Day 1: number analyzed (Participants) | 745 | 738
  B/Victoria, Day 1 | 10.45 [9.6 to 11.4] | 10.36 [9.5 to 11.3]
  B/Victoria, Day 22/50: number analyzed (Participants) | 745 | 738
  B/Victoria, Day 22/50 | 315.52 [287.5 to 346.3] | 138.82 [125.2 to 153.9]
  B/Victoria, Day 181/209: number analyzed (Participants) | 745 | 738
  B/Victoria, Day 181/209 | 65.78 [59.7 to 72.4] | 36.46 [32.9 to 40.4]
Statistical Analysis 1: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); GMT ratio (aQIV/Comparator [TIV/QIV]) for A/H1N1, D22/50 (Pooled Naïve & Non-naïve). An adjusted analysis GMT model (log-transformed postvaccination HI titer = log-transformed prevaccination HI titer+treatment group+ age group, health status+ season + country) was used for analysis; Test type: Superiority — Superiority criterion: The lower bound of the two-sided 95% confidence interval (CI) on the adjusted ratio of GMTs for HI antibody titer exceeds 1; GMT ratio = 1.91, 95% CI 2-sided [1.8 to 2.0]
Statistical Analysis 2: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); GMT ratio (aQIV/Comparator [TIV/QIV]) for A/H1N1, D181/209 (Pooled Naïve & Non-naïve). An adjusted analysis GMT model (log-transformed postvaccination HI titer = log-transformed prevaccination HI titer+treatment group+ age group, health status+ season + country) was used for analysis; Test type: Other; GMT ratio = 1.86, 95% CI 2-sided [1.7 to 2.0]
Statistical Analysis 3: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); GMT ratio (aQIV/Comparator [TIV/QIV]) for A/H3N2, D22/50 (Pooled Naïve & Non-naïve). An adjusted analysis GMT model (log-transformed postvaccination HI titer = log-transformed prevaccination HI titer+treatment group+ age group, health status+ season + country) was used for analysis; Test type: Superiority — Superiority criterion: The lower bound of the two-sided 95% CI on the adjusted ratio of GMTs for HI antibody titer exceeds 1; GMT ratio = 1.71, 95% CI 2-sided [1.6 to 1.8]
Statistical Analysis 4: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); GMT ratio (aQIV/Comparator [TIV/QIV]) for A/H3N2, D181/209 (Pooled Naïve & Non-naïve). An adjusted analysis GMT model (log-transformed postvaccination HI titer = log-transformed prevaccination HI titer+treatment group+ age group, health status+ season + country) was used for analysis; Test type: Other; GMT ratio = 1.57, 95% CI 2-sided [1.4 to 1.7]
Statistical Analysis 5: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); GMT ratio (aQIV/Comparator [TIV/QIV]) for B/YAM, D22/50 (Pooled Naïve & Non-naïve). An adjusted analysis GMT model (log-transformed postvaccination HI titer = log-transformed prevaccination HI titer+treatment group+ age group, health status+ season + country) was used for analysis; Test type: Superiority — [test comment as in outcome 8, analysis 3]; GMT ratio = 2.19, 95% CI 2-sided [2.0 to 2.4]
Statistical Analysis 6: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); GMT ratio (aQIV/Comparator [TIV/QIV]) for B/YAM, D181/209 (Pooled Naïve & Non-naïve). An adjusted analysis GMT model (log-transformed postvaccination HI titer = log-transformed prevaccination HI titer+treatment group+ age group, health status+ season + country) was used for analysis; Test type: Other; GMT ratio = 1.86, 95% CI 2-sided [1.7 to 2.0]
Statistical Analysis 7: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); GMT ratio (aQIV/Comparator [TIV/QIV]) for B/VIC, D22/50 (Pooled Naïve & Non-naïve). An adjusted analysis GMT model (log-transformed postvaccination HI titer = log-transformed prevaccination HI titer+treatment group+ age group, health status+ season + country) was used for analysis; Test type: Superiority — [test comment as in outcome 8, analysis 3]; GMT ratio = 2.27, 95% CI 2-sided [2.0 to 2.6]
Statistical Analysis 8: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); GMT ratio (aQIV/Comparator [TIV/QIV]) for B/VIC, D181/209 (Pooled Naïve & Non-naïve). An adjusted analysis GMT model (log-transformed postvaccination HI titer = log-transformed prevaccination HI titer+treatment group+ age group, health status+ season + country) was used for analysis; Test type: Other; GMT ratio = 1.80, 95% CI 2-sided [1.6 to 2.1]

9. Secondary Outcome: Immunogenicity Endpoint: HI Antibody Responses to aQIV vs TIV/QIV Against Each of the Vaccine Strains in Terms of Geometric Mean Titers (GMTs) in Vaccine Naive Subjects ≥6 to <72 Months of Age
Description: GMTs for vaccine naïve subjects are provided by strain for Day 29 and Day 50; Nonadjuvanted TIV administered in Season 1 and nonadjuvanted QIV administered in Season 2; Homologous strains: A/H1N1=A/California/7/2009 pdm09-like virus, A/H3N2=A/Texas/50/2012, B/ Yamagata=B/Massachusetts/2/2012 and B/Victoria=B/Brisbane/60/2008; For B/Victoria results from Season 2 only are presented for both vaccine groups and used in the vaccine comparison analysis.
Time Frame: Day 29 and Day 50
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- aQIV (≥6 to <72 Months): Vaccine naive subjects ≥6 to <72 months of age who received aQIV
- TIV/QIV (≥6 to <72 Months): Vaccine naive subjects ≥6 to <72 months of age who received TIV/QIV
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 922 | 866
titer
  A/H1N1, Day 29 | 483.55 [395.0 to 591.9] | 172.92 [141.2 to 211.8]
  A/H1N1, Day 50 | 1065.19 [916.0 to 1238.7] | 553.57 [475.5 to 644.4]
  A/H3N2, Day 29 | 742.82 [622.8 to 886.0] | 342.90 [287.4 to 409.1]
  A/H3N2, Day 50 | 1275.18 [1108.8 to 1466.6] | 720.44 [626.0 to 829.1]
  B/Yamagata, Day 29 | 62.73 [51.1 to 77.0] | 31.40 [25.6 to 38.6]
  B/Yamagata, Day 50 | 224.77 [188.6 to 267.9] | 86.91 [72.8 to 103.7]
  B/Victoria, Day 29: number analyzed (Participants) | 411 | 413
  B/Victoria, Day 29 | 81.98 [69.9 to 96.2] | 33.44 [27.9 to 40.1]
  B/Victoria, Day 50: number analyzed (Participants) | 411 | 413
  B/Victoria, Day 50 | 418.16 [376.7 to 464.2] | 160.35 [142.0 to 181.0]

10. Secondary Outcome: Immunogenicity Endpoint: HI Antibody Responses to aQIV vs TIV/QIV Against Each of the Vaccine Strains in Terms GMT and GMT Ratios at 21 Days After Last Vaccination in Healthy vs High Risk Subjects ≥6 to <72 Months of Age
Description: HI GMT was assessed on Day 1 and Day 50 for vaccine naïve healthy vs high risk subjects; and HI GMT were assessed on Day 1 and Day 22 for vaccine non-naïve healthy vs high risk subjects; pooled GMT values across both naïve and non-naïve subjects are provided for Day 22/50 (ie, 21 days after last vaccination) assessments.
Time Frame: Baseline (Day 1) and 21 days after the last vaccination (Day 50 for vaccine naive subjects; Day 22 for vaccine non-naïve subjects)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- aQIV (≥6 to <72 Months) - Healthy: Healthy subjects ≥6 to <72 months of age who received aQIV
- aQIV (≥6 to <72 Months) - High Risk: High risk subjects ≥6 to <72 months of age who received aQIV
- TIV/QIV (≥6 to <72 Months) - Healthy: Healthy subjects ≥6 to <72 months of age who received TIV/QIV
- TIV/QIV (≥6 to <72 Months) - High Risk: High risk subjects ≥6 to <72 months of age who received TIV/QIV
Arm/Group | aQIV (≥6 to <72 Months) - Healthy | aQIV (≥6 to <72 Months) - High Risk | TIV/QIV (≥6 to <72 Months) - Healthy | TIV/QIV (≥6 to <72 Months) - High Risk
Number analyzed (Participants) | 1208 | 273 | 1171 | 234
titer
  A/H1N1, Day 1 | 35.34 [26.4 to 47.2] | 48.29 [34.7 to 67.2] | 31.64 [23.3 to 42.9] | 45.12 [31.9 to 63.8]
  A/H1N1, Day 22/50 | 988.65 [863.68 to 1131.6] | 906.86 [777.8 to 1057.3] | 563.87 [471.8 to 674.0] | 533.71 [436.8 to 652.2]
  A/H3N2, Day 1 | 76.80 [56.3 to 104.8] | 104.07 [73.0 to 148.3] | 55.08 [40.1 to 75.8] | 59.89 [41.7 to 85.9]
  A/H3N2, Day 22/50 | 1159.57 [1017.2 to 1321.9] | 1179.55 [1015.7 to 1369.9] | 693.27 [589.4 to 815.4] | 680.08 [566.6 to 816.2]
  B/YAM, Day 1 | 9.95 [8.5 to 11.7] | 11.72 [9.7 to 14.1] | 8.76 [7.4 to 10.4] | 10.18 [8.4 to 12.4]
  B/YAM, Day 22/50 | 203.14 [169.6 to 243.4] | 198.58 [161.7 to 243.9] | 94.76 [77.6 to 115.8] | 89.59 [71.5 to 112.1]
  B/VIC, Day 1 | 10.87 [9.1 to 12.9] | 10.51 [8.6 to 12.8] | 8.17 [6.6 to 10.1] | 9.03 [7.1 to 11.5]
  B/VIC, Day 22/50 | 323.42 [264.0 to 396.2] | 298.20 [236.7 to 375.7] | 151.17 [120.3 to 189.9] | 138.94 [107.3 to 179.9]
Statistical Analysis 1: Comparison: aQIV (≥6 to <72 Months) - Healthy vs aQIV (≥6 to <72 Months) - High Risk; aQIV GMT ratio (High risk/Healthy) for A/H1N1 at D22/50 (Pooled Naïve & Non-naïve); Test type: Other; GMT ratio = 0.92, 95% CI 2-sided [0.8 to 1.0]
Statistical Analysis 2: Comparison: aQIV (≥6 to <72 Months) - Healthy vs aQIV (≥6 to <72 Months) - High Risk; aQIV GMT ratio (High risk/Healthy) for A/H3N2 at D22/50 (Pooled Naïve & Non-naïve); Test type: Other; GMT ratio = 1.02, 95% CI 2-sided [0.9 to 1.1]
Statistical Analysis 3: Comparison: aQIV (≥6 to <72 Months) - Healthy vs aQIV (≥6 to <72 Months) - High Risk; aQIV GMT ratio (High risk/Healthy) for B/YAM at D22/50 (Pooled Naïve & Non-naïve); Test type: Other; GMT ratio = 0.98, 95% CI 2-sided [0.8 to 1.1]
Statistical Analysis 4: Comparison: aQIV (≥6 to <72 Months) - Healthy vs aQIV (≥6 to <72 Months) - High Risk; aQIV GMT ratio (High risk/Healthy) for B/VIC at D22/50 (Pooled Naïve & Non-naïve); Test type: Other; GMT ratio = 0.92, 95% CI 2-sided [0.8 to 1.1]
Statistical Analysis 5: Comparison: TIV/QIV (≥6 to <72 Months) - Healthy vs TIV/QIV (≥6 to <72 Months) - High Risk; TIV/QIV GMT ratio (High risk/Healthy) for A/H1N1 at D22/50 (Pooled Naïve & Non-naïve); Test type: Other; GMT ratio = 0.95, 95% CI 2-sided [0.8 to 1.1]
Statistical Analysis 6: Comparison: TIV/QIV (≥6 to <72 Months) - Healthy vs TIV/QIV (≥6 to <72 Months) - High Risk; TIV/QIV GMT ratio (High risk/Healthy) for A/H3N2 at D22/50 (Pooled Naïve & Non-naïve); Test type: Other; GMT ratio = 0.98, 95% CI 2-sided [0.8 to 1.1]
Statistical Analysis 7: Comparison: TIV/QIV (≥6 to <72 Months) - Healthy vs TIV/QIV (≥6 to <72 Months) - High Risk; TIV/QIV GMT ratio (High risk/Healthy) for B/YAM at D22/50 (Pooled Naïve & Non-naïve); Test type: Other; GMT ratio = 0.95, 95% CI 2-sided [0.8 to 1.1]
Statistical Analysis 8: Comparison: TIV/QIV (≥6 to <72 Months) - Healthy vs TIV/QIV (≥6 to <72 Months) - High Risk; TIV/QIV GMT ratio (High risk/Healthy) for B/VIC at D22/50 (Pooled Naïve & Non-naïve); Test type: Other; GMT ratio = 0.92, 95% CI 2-sided [0.7 to 1.2]

11. Secondary Outcome: Immunogenicity Endpoint: HI Antibody Responses to aQIV vs TIV/QIV Against Each of the Vaccine Strains in Terms of Geometric Mean Ratios (GMR) in Subjects ≥6 to <72 Months of Age
Description: The fold-increase in HI antibodies in response to vaccination was assessed as the GMR between all post-vaccination titers (ie, Day 29, 50, 209 for vaccine naïve subjects; Day 22, 181 for vaccine non-naïve subjects) and the baseline (Day 1) titer. Assessed GMRs thus correspond to Day 29/Day 1, Day 50/Day 1, and Day 209/Day 1 for vaccine naïve subjects and Day 22/Day 1 and Day 181/Day 1 for vaccine non-naïve subjects. Pooled GMR values across both naïve and non-naïve subjects are provided for Day (22/50)/Day 1 (ie, 21 days after last vaccination) and Day (181/209)/Day 1 (ie, 180 days after last vaccination); Nonadjuvanted TIV administered in Season 1 and nonadjuvanted QIV administered in Season 2; Homologous strains: A/H1N1=A/California/7/2009 pdm09-like virus, A/H3N2=A/Texas/50/2012, B/Yamagata=B/Massachusetts/2/2012 and B/Victoria=B/Brisbane/60/2008; For B/Victoria results from Season 2 only are presented for both vaccine groups and used in the vaccine comparison analysis.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 1481 | 1405
ratio
  A/H1N1, Day 22/50:Day 1 | 24.96 [22.3 to 28.0] | 13.09 [11.7 to 14.7]
  A/H3N2, Day 22/50:Day 1 | 21.68 [19.5 to 24.1] | 12.67 [11.4 to 14.1]
  B/Yamagata, Day 22/50:Day 1 | 18.08 [15.7 to 20.8] | 8.25 [7.2 to 9.5]
  B/Victoria, Day 22/50/Day 1: number analyzed (Participants) | 745 | 738
  B/Victoria, Day 22/50/Day 1 | 29.70 [26.9 to 32.7] | 13.28 [12.0 to 14.7]
  A/H1N1, Day 181/209:Day 1 | 8.57 [7.6 to 9.7] | 4.62 [4.1 to 5.2]
  A/H3N2, Day 181/209:Day 1 | 8.64 [7.6 to 9.8] | 5.49 [4.8 to 6.2]
  B/Yamagata Day 181/209:Day 1 | 4.38 [3.9 to 5.0] | 2.36 [2.1 to 2.7]
  B/Victoria, Day 181/209/Day 1: number analyzed (Participants) | 745 | 738
  B/Victoria, Day 181/209/Day 1 | 6.28 [5.7 to 6.9] | 3.56 [3.3 to 3.9]

12. Secondary Outcome: Immunogenicity Endpoint: HI Antibody Responses to aQIV vs TIV/QIV Against Each of the Vaccine Strains in Terms of Seroconversion (SC) Rates and Difference in SC Rates at 21 Days in Subjects ≥6 to <72 Months of Age
Description: SC rates were assessed on Day 1 and Day 50 (ie, 21 days after two vaccinations) for vaccine naïve subjects; and on Day 1 and Day 22 (ie, 21 days after one vaccination) for vaccine non-naïve subjects; values pooled across naive and non-naive subjects are provided. Seroconversion is defined as HI ≥ 1:40 for subjects negative at baseline (ie, HI titer<1:10); or a minimum 4-fold increase in HI titer for subjects positive at baseline (ie, HI titer ≥ 1:10); Nonadjuvanted TIV administered in Season 1 and nonadjuvanted QIV administered in Season 2; Homologous strain: A/H1N1=A/California/7/2009 pdm09-like virus, A/H3N2=A/Texas/50/2012, B/Yamagata=B/Massachusetts/2/2012 and B/Victoria=B/Brisbane/60/2008; For B/Victoria results from Season 2 only are presented for both vaccine groups and used in the vaccine.
  comparison analysis (N=745 for aQIV, N=738 for comparator).
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 1481 | 1405
percentage of subjects
  A/H1N1 | 81.9 [79.7 to 83.9] | 73.7 [71.2 to 76.1]
  A/H3N2 | 78.4 [76.1 to 80.6] | 73.2 [70.7 to 75.6]
  B/Yamagata | 86.0 [84.1 to 87.8] | 64.7 [62.1 to 67.3]
  B/Victoria: number analyzed (Participants) | 745 | 738
  B/Victoria | 91.0 [88.8 to 93.0] | 77.4 [74.2 to 80.3]
Statistical Analysis 1: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Seroconversion difference (aQIV - Comparator [TIV/QIV]) for A/H1N1; Test type: Superiority — Superiority criterion: The lower bound of the two-sided 95% CI on the unadjusted difference of percentages of subjects seroconverted for HI antibody exceeds 0%; Seroconversion difference = 8.2, 95% CI 2-sided [5.0 to 11.3]
Statistical Analysis 2: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Seroconversion difference (aQIV - Comparator [TIV/QIV]) for A/H3N2; Test type: Superiority — [test comment as in outcome 12, analysis 1]; Seroconversion difference = 5.2, 95% CI 2-sided [1.9 to 8.4]
Statistical Analysis 3: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Seroconversion difference (aQIV - Comparator [TIV/QIV]) for B/YAM; Test type: Superiority; Seroconversion difference = 21.3, 95% CI 2-sided [18.1 to 24.5]
Statistical Analysis 4: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Seroconversion difference (aQIV - Comparator [TIV/QIV]) for B/VIC; Test type: Superiority — [test comment as in outcome 12, analysis 1]; Seroconversion difference = 13.6, 95% CI 2-sided [10.0 to 17.3]

13. Secondary Outcome: Immunogenicity Endpoint: HI Antibody Responses to aQIV vs TIV/QIV Against Each of the Vaccine Strains in Terms of Percentage of Subjects With HI Titer ≥ 1:40 and Percentage Differences at 180 Days After Last Vaccination in Subjects ≥6 to <72 Months of Age
Description: Antibody response was assessed as the percentage of subjects with HI titer of ≥1:40 at 180 days after last vaccination (ie, Day 209 for vaccine naïve subjects and Day 181 for vaccine non-naïve subjects). Results were then pooled across both vaccine naïve and non-naïve subjects. Homologous strains: A/H1N1=A/California/7/2009 pdm09-like virus, A/H3N2=A/Texas/50/2012, B/Yamagata=B/Massachusetts/2/2012 and B/Victoria=B/Brisbane/60/2008; B/Victoria results from Season 1 and Season 2 (aQIV) and Season 2 (comparator) are presented.
Time Frame: Baseline (Day 1) and 180 days after the last vaccination (Day 209 for vaccine naive subjects; Day 181 for vaccine non-naïve subjects)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 1481 | 1405
percentage of subjects
  A/H1N1 | 97.1 [96.0 to 98.0] | 85.6 [83.6 to 87.5]
  A/H3N2 | 98.1 [97.1 to 98.7] | 90.2 [88.4 to 91.8]
  B/Yamagata | 66.6 [63.9 to 69.2] | 44.7 [41.9 to 47.5]
  B/Victoria: number analyzed (Participants) | 745 | 738
  B/Victoria | 74.0 [70.6 to 77.2] | 53.1 [49.4 to 56.9]
Statistical Analysis 1: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI titers ≥ 1:40 (aQIV - Comparator [TIV/QIV]) for A/H1N1; Test type: Other; Mean Difference (Final Values) = 11.5, 95% CI 2-sided [9.4 to 13.7]
Statistical Analysis 2: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI titers ≥ 1:40 (aQIV - Comparator [TIV/QIV]) for A/H3N2; Test type: Other; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [6.1 to 9.7]
Statistical Analysis 3: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI titers ≥ 1:40 (aQIV - Comparator [TIV/QIV]) for B/YAM; Test type: Other; Mean Difference (Final Values) = 21.9, 95% CI 2-sided [18.1 to 25.6]
Statistical Analysis 4: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI titers ≥ 1:40 (aQIV - Comparator [TIV/QIV]) for B/VIC; Test type: Other; Mean Difference (Final Values) = 20.9, 95% CI 2-sided [15.9 to 25.7]

14. Secondary Outcome: Immunogenicity Endpoint: HI Antibody Responses to aQIV vs TIV/QIV Against Each of the Vaccine Strains in Terms of Percentage of Subjects With HI Titers ≥1:110, ≥1:151, ≥1:215, ≥1:330, and ≥1:629 in Subjects ≥6 to <72 Months of Age
Description: Antibody response was assessed as the percentage of subjects and differences of percentage of subjects with HI titers of ≥1:110, ≥1:151, ≥1:215, ≥1:330, and ≥1:629 at 21 days after last vaccination (ie, Day 50 for vaccine naïve subjects and Day 22 for vaccine non-naïve subjects). Results were then pooled across both vaccine naïve and non-naïve subjects. Homologous strains: A/H1N1=A/California/7/2009 pdm09-like virus, A/H3N2=A/Texas/50/2012, B/Yamagata=B/Massachusetts/2/2012 and B/Victoria=B/Brisbane/60/2008; B/Victoria results from Season 1 and Season 2 (aQIV) and Season 2 (comparator) are presented.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 1481 | 1405
percentage of subjects
  HI Titers ≥1:110, A/H1N1, Day 22/50 | 97.3 [96.3 to 98.1] | 89.5 [87.7 to 91.1]
  HI Titers ≥1:151, A/H1N1, Day 22/50 | 96.5 [95.4 to 97.5] | 86.8 [84.8 to 88.6]
  HI Titers ≥1:215, A/H1N1, Day 22/50 | 94.0 [92.6 to 95.2] | 77.9 [75.5 to 80.1]
  HI Titers ≥1:330, A/H1N1, Day 22/50 | 83.8 [81.8 to 85.8] | 60.7 [58.0 to 63.4]
  HI Titers ≥1:629, A/H1N1, Day 22/50 | 76.2 [73.9 to 78.5] | 52.1 [49.4 to 54.8]
  HI Titers ≥1:110, A/H3N2, Day 22/50 | 99.0 [98.3 to 99.4] | 93.0 [91.5 to 94.4]
  HI Titers ≥1:151, A/H3N2, Day 22/50 | 98.4 [97.6 to 99.0] | 90.6 [88.9 to 92.1]
  HI Titers ≥1:215, A/H3N2, Day 22/50 | 96.5 [95.4 to 97.4] | 84.8 [82.7 to 86.7]
  HI Titers ≥1:330, A/H3N2, Day 22/50 | 89.4 [87.7 to 91.0] | 70.4 [67.8 to 72.9]
  HI Titers ≥1:629, A/H3N2, Day 22/50 | 84.2 [82.2 to 86.1] | 63.1 [60.4 to 65.7]
  HI Titers ≥1:110, B/YAM, Day 22/50 | 69.4 [66.9 to 71.8] | 40.6 [38.0 to 43.3]
  HI Titers ≥1:151, B/YAM, Day 22/50 | 60.7 [58.1 to 63.3] | 34.4 [31.9 to 37.1]
  HI Titers ≥1:215, B/YAM, Day 22/50 | 45.6 [42.9 to 48.3] | 23.8 [21.5 to 26.2]
  HI Titers ≥1:330, B/YAM, Day 22/50 | 24.9 [22.6 to 27.3] | 13.3 [11.5 to 15.3]
  HI Titers ≥1:629, B/YAM, Day 22/50 | 16.2 [14.3 to 18.3] | 9.4 [7.9 to 11.1]
  HI Titers ≥1:110, B/VIC, Day 22/50: number analyzed (Participants) | 1481 | 738
  HI Titers ≥1:110, B/VIC, Day 22/50 | 78.3 [76.0 to 80.4] | 58.1 [54.5 to 61.7]
  HI Titers ≥1:151, B/VIC, Day 22/50: number analyzed (Participants) | 1481 | 738
  HI Titers ≥1:151, B/VIC, Day 22/50 | 73.5 [71.1 to 75.8] | 52.4 [48.8 to 56.1]
  HI Titers ≥1:215, B/VIC, Day 22/50: number analyzed (Participants) | 1481 | 738
  HI Titers ≥1:215, B/VIC, Day 22/50 | 62.3 [59.7 to 64.9] | 38.6 [35.1 to 42.2]
  HI Titers ≥1:330, B/VIC, Day 22/50: number analyzed (Participants) | 1481 | 738
  HI Titers ≥1:330, B/VIC, Day 22/50 | 41.7 [39.1 to 44.4] | 21.8 [18.9 to 25.0]
  HI Titers ≥1:629, B/VIC, Day 22/50: number analyzed (Participants) | 1481 | 738
  HI Titers ≥1:629, B/VIC, Day 22/50 | 31.9 [29.4 to 34.4] | 16.9 [14.3 to 19.8]
Statistical Analysis 1: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI titers ≥ 1:110 for A/H1N1 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [5.9 to 9.7]
Statistical Analysis 2: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:151 for A/H1N1 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 9.8, 95% CI 2-sided [7.8 to 11.9]
Statistical Analysis 3: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:215 for A/H1N1 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 16.1, 95% CI 2-sided [13.5 to 18.7]
Statistical Analysis 4: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:330 for A/H1N1 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 23.1, 95% CI 2-sided [19.8 to 26.4]
Statistical Analysis 5: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:629 for A/H1N1 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 24.1, 95% CI 2-sided [20.6 to 27.6]
Statistical Analysis 6: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:110 for A/H3N2 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [4.5 to 7.5]
Statistical Analysis 7: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:151 for A/H3N2 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [6.1 to 9.6]
Statistical Analysis 8: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:215 for A/H3N2 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 11.7, 95% CI 2-sided [9.6 to 13.9]
Statistical Analysis 9: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:330 for A/H3N2 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 19.0, 95% CI 2-sided [16.1 to 22.0]
Statistical Analysis 10: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:629 for A/H3N2 (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 21.1, 95% CI 2-sided [17.8 to 24.3]
Statistical Analysis 11: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:110 for B/YAM (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 28.8, 95% CI 2-sided [25.1 to 32.3]
Statistical Analysis 12: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:151 for B/YAM (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 26.3, 95% CI 2-sided [22.6 to 29.9]
Statistical Analysis 13: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:215 for B/YAM (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 21.8, 95% CI 2-sided [18.3 to 25.3]
Statistical Analysis 14: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:330 for B/YAM (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 11.6, 95% CI 2-sided [8.6 to 14.5]
Statistical Analysis 15: Comparison: aQIV (≥6 to <72 Months) vs TIV/QIV (≥6 to <72 Months); Difference in HI Titers ≥ 1:629 for B/YAM (aQIV - Comparator [TIV/QIV]) at Day 22/50; Test type: Other; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [4.3 to 9.4]

15. Secondary Outcome: Immunogenicity Endpoint: Hemagglutination Inhibition (HI) Antibody Responses to aQIV vs TIV/QIV Against Heterologous Strains in Terms of Geometric Mean Titers (GMTs) in Subjects ≥6 to <72 Months of Age
Description: HI GMT was assessed 21 days after last vaccination (Day 50 for vaccine naïve subjects and Day 22 for vaccine non-naive subjects) pooled GMT values across both naïve and non-naïve subjects are provided for the Day 22/50 (ie, 21 days after last vaccination); Heterologous strains: H1N1=A/Brisbane/59/2007- like; H3N2 =A/Hong Kong/4801/2014; B/Yamagata=B/Phuket/3073/2013-like; B Victoria=B/Malaysia/2506/2004; For B/Victoria results from Season 2 only are presented for both vaccine groups.
Time Frame: 21 days after the last vaccination (Day 50 for vaccine naive subjects; Day 22 for vaccine non-naïve subjects)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 297 | 295
titer
  A/H1N1, D22/50 | 7.46 [6.3 to 8.9] | 6.52 [5.5 to 7.8]
  A/H3N2, D22/50 | 576.84 [407.4 to 816.7] | 297.70 [209.0 to 424.1]
  B/Yamagata, Day 22/50 | 145.89 [98.3 to 216.6] | 67.24 [45.0 to 100.5]
  B/Victoria, Day 22/50: number analyzed (Participants) | 141 | 158
  B/Victoria, Day 22/50 | 186.65 [157.3 to 221.5] | 88.09 [73.0 to 106.3]

16. Secondary Outcome: Immunogenicity Endpoint: HI Antibody Responses to aQIV vs TIV/QIV Heterologous Strains in Terms of Seroconversion (SC) Rates in Subjects ≥6 to <72 Months of Age
Description: SC rates were assessed on Day 50 (ie, 21 days after two vaccinations) for vaccine naïve subjects; and on Day 22 (ie, 21 days after one vaccination) for vaccine non-naïve subjects; values pooled across naive and non-naive subjects are provided. Seroconversion is defined as HI ≥ 1:40 for subjects negative at baseline (ie, HI titer<1:10); or a minimum 4-fold increase in HI titer for subjects positive at baseline (ie, HI titer ≥ 1:10); Heterologous strains include: H1N1=A/Brisbane/59/2007- like; H3N2 =A/Hong Kong/4801/2014; B/Yamagata=B/Phuket/3073/2013- like; B Victoria=B/Malaysia/2506/2004; For B/Victoria results from Season 2 only are presented for both vaccine groups
Time Frame: 21 days after the last vaccination (Day 50 for vaccine naive subjects; Day 22 for vaccine non-naïve subjects)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 297 | 295
percentage of subjects
  A/H1N1 | 2.7 [1.2 to 5.3] | 1.4 [0.4 to 3.5]
  A/H3N2 | 86.0 [81.4 to 89.7] | 73.4 [68.0 to 78.4]
  B/Yamagata | 82.7 [77.9 to 86.8] | 59.9 [54.1 to 65.6]
  B/Victoria: number analyzed (Participants) | 140 | 157
  B/Victoria | 90.7 [84.6 to 95.0] | 75.8 [68.3 to 82.3]

17. Secondary Outcome: Immunogenicity Endpoint: HI Antibody Responses to aQIV vs TIV/QIV Against Heterologous Strains in Terms of Percentage of Subjects With HI Titer ≥ 1:40 in Subjects ≥6 to <72 Months of Age
Description: Antibody persistence was assessed as the percentage of subjects with HI titer of ≥1:40 at 21 days after last vaccination (ie, Day 50 for vaccine naïve subjects and Day 22 for vaccine non-naïve subjects). Results were then pooled across both vaccine naïve and non-naïve subjects; Heterologous strains: H1N1=A/Brisbane/59/2007- like; H3N2 =A/Hong Kong/4801/2014; B/Yamagata=B/Phuket/3073/2013- like; B Victoria=B/Malaysia/2506/2004; For B/Victoria results from Season 2 only are presented for both vaccine groups.
Time Frame: 21 days after the last vaccination (Day 50 for vaccine naive subjects; Day 22 for vaccine non-naïve subjects)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 297 | 295
percentage of subjects
  A/H1N1 | 6.1 [3.7 to 9.5] | 3.4 [1.7 to 6.2]
  A/H3N2 | 99.3 [97.5 to 99.9] | 93.1 [89.5 to 95.7]
  B/Yamagata | 88.8 [84.6 to 92.2] | 68.2 [62.5 to 73.5]
  B/Victoria | 95.7 [90.9 to 98.4] | 83.4 [76.7 to 88.9]

18. Secondary Outcome: Safety Endpoint: Number of Subjects With Solicited Local and Systemic AEs
Description: Subjects ≥6 to <72 months of age reporting solicited local and systemic reactions, day 1 to day 7 after vaccination with either aQIV or TIV/QIV.
Time Frame: 7 days following each vaccination
Population: The Solicited Safety Set consisting of all subjects who received a study vaccination and had any assessment of local and systemic reactions and/or assessment of any use of analgesics/antipyretics was used for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 5138 | 5056
Participants
  Any | 3748 | 3242
  Local | 2651 | 2188
  Systemic | 2714 | 2174
  Others | 1536 | 907

19. Secondary Outcome: Safety Endpoint: Number of Subjects With Unsolicited AEs, SAEs, AEs Leading to Withdrawal From the Study or Study Vaccination, NOCDs and AESIs
Description: Safety was assessed in terms of number of subjects ≥6 to <72 months of age reporting unsolicited reactions (Day 1 to Day 50 for vaccine naïve subjects and from Day 1 to Day 22 for vaccine non-naïve subjects); Serious Adverse Events (SAEs), AEs leading to New Onset of Chronic Diseases,(NOCD), Adverse Events of Special Interests (AESI), AEs leading to withdrawal from the study or study vaccination after vaccination with either aQIV or TIV/QIV were collected up to 12 months after last vaccination.
Time Frame: Day 1 though Day 366 (vaccine non-naive)/Day 390 (vaccine naive)
Population: The Unsolicited Safety Set consisting of all subjects who received a study vaccination and had any AE assessments was used for analysis (ie, a subject did not have to have an AE to be included in this population).
Measure: Count of Participants; unit: Participants
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
Number analyzed (Participants) | 5243 | 5161
Participants
  Any unsolicited AEs | 3576 | 3543
  Possibly or probably related unsolicited AEs | 686 | 533
  SAEs | 234 | 230
  Possibly or probably related SAEs | 6 | 1
  AEs with an outcome of death | 1 | 3
  AEs leading to withdrawal | 10 | 9
  AEs leading to NOCD | 87 | 96
  AESIs | 5 | 4

20. Secondary Outcome: Healthcare Utilization and Health Economic Endpoints: Number of Days of Daycare, School or Preschool Missed by Subjects Associated With RT-PCR-confirmed Influenza
Time Frame: within a window of 14 days after influenza-like illness (ILI)-onset
Population: Full Analysis Set Health Economic Outcomes (Season 2): This analysis set includes all subjects in the Enrolled Set in Season 2 who: actually received a study vaccination and provided efficacy data and Health Economic data collected within 14 days of ILI-onset; and had a first-occurrence RT-PCR-confirmed influenza as included in the primary efficacy objective.
Measure: Mean (Standard Deviation); unit: Number of days
Groups:
- aQIV (≥6 to <72 Months): Subjects ≥6 to <72 months of age who received aQIV in Season 2
- QIV (≥6 to <72 Months): Subjects ≥6 to <72 months of age who received QIV in Season 2
Arm/Group | aQIV (≥6 to <72 Months) | QIV (≥6 to <72 Months)
Number analyzed (Participants) | 255 | 250
Number of days | 2.1 (2.43) | 2.2 (2.48)

21. Secondary Outcome: Healthcare Utilization and Health Economic Endpoint: Number of Medical Visit for Respiratory Illness Associated With RT-PCR-confirmed Influenza
Time Frame: within a window of 14 days after ILI-onset
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | aQIV (≥6 to <72 Months) | QIV (≥6 to <72 Months)
Number analyzed (Participants) | 255 | 250
Number of visits | 1.0 (0.84) | 1.0 (0.74)

22. Secondary Outcome: Healthcare Utilization and Health Economic Endpoint: Number of Employment Days Missed by Parent(s)/Guardian(s) of Subjects With RT-PCR-confirmed Influenza
Time Frame: within a window of 14 days after ILI-onset
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | aQIV (≥6 to <72 Months) | QIV (≥6 to <72 Months)
Number analyzed (Participants) | 255 | 250
Number of days | 1.0 (1.68) | 1.0 (1.88)

23. Secondary Outcome: Healthcare Utilization and Health Economic Endpoint: First-occurrence of RT-PCR-confirmed Moderate-to-severe Influenza Cases as Per Prespecified Criteria in Subjects ≥6 to <72 Months of Age in Season 2.
Time Frame: as for outcome 1
Population: Full Analysis Set Health Economic Outcomes (Season 2)
Measure: Number; unit: Number of cases
Arm/Group | aQIV (≥6 to <72 Months) | QIV (≥6 to <72 Months)
Number analyzed (Participants) | 255 | 250
Number of cases
  Any Strain | 34 | 32
  A/H1N1 | 0 | 1
  A/H3N2 | 27 | 29
  B/Yamagata | 4 | 2
  B/Victoria | 3 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 366 (for vaccine non-naive subjects) and Day 1 to Day 390 (for vaccine naive subjects). AEs are reported for the aQIV arm and the TIV/QIV arm. Although randomization was stratified by vaccination influenza history (naive vs non-naive), which determined the number of doses of vaccine a subject received, the intention was to report the safety results for each arm as a whole.
Description: SAEs: Day 1 to Day 366 for vaccine non-naive and Day 1 to Day 390 for vaccine naive subjects.
  Non-serious AEs: solicited AEs: Day 1 to Day 7 after each vaccination; and unsolicited AEs: Day 1 to Day 366 for vaccine non-naive and Day 1 to Day 390 for vaccine naive subjects.
  All-cause mortality and non-serious AEs are reported for the Overall Safety Set (all subjects in the Solicited Safety Set and/or in the Unsolicited Safety Set). SAEs are reported for the Unsolicited Safety Set.
Arm/Group | aQIV (≥6 to <72 Months) | TIV/QIV (≥6 to <72 Months)
All-Cause Mortality (participants affected / at risk) | 1/5339 | 3/5272
Serious Adverse Events (participants affected / at risk) | 234/5243 | 230/5161
Other Adverse Events (participants affected / at risk) | 4627/5339 | 4430/5272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (≥6 to <72 Months) (N=5243) | TIV/QIV (≥6 to <72 Months) (N=5161)
Kawasaki's disease (Vascular disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Type I hypersensitivity (Immune system disorders) | 1 | 0
Influenza like illness (General disorders) | 7 | 8
Pyrexia (General disorders) | 1 | 6
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Accidental exposure to product (Injury, poisoning and procedural complications) | 2 | 1
Animal bite (Injury, poisoning and procedural complications) | 24 | 19
Animal scratch (Injury, poisoning and procedural complications) | 2 | 3
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Chemical burn of gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 1
Foreign body (Injury, poisoning and procedural complications) | 1 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 2
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 1
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 1
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Autism (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Encephalitis autoimmune (Nervous system disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 13 | 7
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 1
Status epilepticus (Nervous system disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 5 | 5
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 2
Device malfunction (Product Issues) | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperaldosteronism (Endocrine disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 15 | 11
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess jaw (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 2
Amoebiasis (Infections and infestations) | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 7 | 1
Bronchitis (Infections and infestations) | 12 | 13
Cellulitis (Infections and infestations) | 5 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Cholera (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 1
Croup infectious (Infections and infestations) | 3 | 2
Dengue fever (Infections and infestations) | 9 | 9
Diarrhoea infectious (Infections and infestations) | 0 | 2
Exanthema subitum (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastritis viral (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 23 | 23
Gastroenteritis rotavirus (Infections and infestations) | 0 | 5
Gastroenteritis salmonella (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 3 | 4
Groin abscess (Infections and infestations) | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 2 | 4
Herpangina (Infections and infestations) | 5 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 1
Laryngitis viral (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Mycoplasma infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 1
Otitis media acute (Infections and infestations) | 2 | 0
Periorbital cellulitis (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 4 | 7
Pharyngotonsillitis (Infections and infestations) | 3 | 3
Pneumonia (Infections and infestations) | 38 | 28
Pneumonia adenoviral (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 3 | 2
Pneumonia viral (Infections and infestations) | 4 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 3 | 3
Respiratory tract infection (Infections and infestations) | 1 | 2
Rhinitis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal scalded skin syndrome (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 3 | 1
Tonsillitis (Infections and infestations) | 5 | 3
Tooth abscess (Infections and infestations) | 0 | 1
Typhoid fever (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 3 | 7
Viral diarrhoea (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 4 | 3
Viral pharyngitis (Infections and infestations) | 1 | 0
Viral rash (Infections and infestations) | 1 | 1
Viral sinusitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Injection site inflammation (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aQIV (≥6 to <72 Months) (N=5339) | TIV/QIV (≥6 to <72 Months) (N=5272)
Cough (Respiratory, thoracic and mediastinal disorders) | 305 | 312
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 206 | 225
Somnolence (Nervous system disorders) | 1366 | 1107
Influenza like illness (General disorders) | 2690 | 2664
Injection site pain (General disorders) | 2360 | 1861
Injection site erythema (General disorders) | 1226 | 1031
Pyrexia (General disorders) | 1178 | 778
Injection site induration (General disorders) | 804 | 576
Injection site haemorrhage (General disorders) | 407 | 374
Chills (General disorders) | 356 | 210
Irritability (Psychiatric disorders) | 1441 | 1204
Eating disorder (Psychiatric disorders) | 1163 | 898
Diarrhoea (Gastrointestinal disorders) | 701 | 677
Vomiting (Gastrointestinal disorders) | 634 | 516
Upper respiratory tract infection (Infections and infestations) | 722 | 724
Nasopharyngitis (Infections and infestations) | 387 | 365
Otitis media (Infections and infestations) | 375 | 352
Pneumonia (Infections and infestations) | 218 | 241
Rhinitis (Infections and infestations) | 215 | 221
Bronchitis (Infections and infestations) | 186 | 201
Gastroenteritis (Infections and infestations) | 156 | 139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less